CLINICAL TRIAL: NCT00330590
Title: Central Venous Access Catheter Placement by Interventional Radiologists Using the Sonic Flashlight for Real Time Ultrasound Guidance
Brief Title: Central Venous Access Catheter Placement Using the Sonic Flashlight
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Other Study IDs: 0512052
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Catheterization, Central Venous
Keywords: Central Venous; Ultrasonography; Catheterization

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The investigators have developed a new device for guiding invasive procedures with ultrasound (US), which they call the sonic flashlight (SF). They attach a half-silvered mirror and a small flat-panel monitor directly to an ultrasound transducer to project a virtual image of the US scan into its actual location within the patient. This permits the operator to guide a needle through the skin by aiming directly at the image, using natural hand-eye coordination rather than looking away from the patient at a conventional display. The device requires no tracking or head-mounted apparatus, and provides an intuitive merger of the visual exterior of the patient with an in situ ultrasound image, which can be simultaneously viewed by others assisting the operator. The investigators believe the SF will increase the accuracy, safety, and speed for a wide variety of invasive procedures, and will require less extensive training than conventional US displays.

Given the wide variety of procedures for which the SF could be used, the investigators have narrowed their focus to applying it to a single application: vascular access. They have demonstrated clinically that the SF can be used successfully to guide the placement of the peripherally inserted central catheter (PICC) lines. The research proposed here will expand this application to include the insertion of other central venous access (CVA) lines through the internal jugular vein, subclavian vein, and femoral vein. The historical approach to CVA line placements has involved the physical exam and identification of visible landmarks. With the introduction and common usage of ultrasound, it has become routine to use ultrasound guidance.

Much of the difficulty in learning conventional ultrasound (CUS) guided procedures stems from the displaced sense of hand-eye coordination that occurs when the operator looks away from the operating field to see the ultrasound display. The SF directly addresses many of these issues and therefore the investigators believe that it is well suited for this application. They have already shown that novice US users learn vascular access procedures in training phantoms more quickly using the SF than CUS. They have also shown that intravenous (IV) team nurses already proficient in CUS guided PICC lines perform vascular access in training phantoms more quickly using the SF than CUS guidance. Finally, as mentioned earlier, the investigators have shown that the SF can be used successfully to guide the placement of PICC lines. This study will test the hypothesis that the SF will successfully facilitate catheter placement in the subclavian, femoral, and internal jugular veins demonstrating equal vasculature visualization as conventional ultrasound.

DETAILED DESCRIPTION:
We have developed a new device for guiding invasive procedures with ultrasound (US), which we call the Sonic Flashlight (SF). We attach a half-silvered mirror and a small flat-panel monitor directly to an ultrasound transducer to project a virtual image of the US scan into its actual location within the patient. This permits the operator to guide a needle through the skin by aiming directly at the image, using natural hand-eye coordination rather than looking away from the patient at a conventional display. The device requires no tracking or head-mounted apparatus, and provides an intuitive merger of the visual exterior of the patient with an in situ ultrasound image, which can be simultaneously viewed by others assisting the operator. We believe the SF will increase accuracy, safety, and speed, for a wide variety of invasive procedures, and will require less extensive training than conventional US displays.

Given the wide variety of procedures for which the SF could be used, we have narrowed our focus to applying it to a single application: vascular access. We have demonstrated clinically that the SF can be used successfully to guide the placement of the Peripherally Inserted Central Catheter (PICC) lines. The research proposed here will expand this application to include the insertion of other Central Venous Access (CVA) lines through the internal jugular vein, subclavian vein, and femoral vein. The historical approach to CVA line placements has involved the physical exam and identification of visible landmarks. With the introduction and common usage of ultrasound, it has become routine to use ultrasound guidance.

Much of the difficulty in learning conventional ultrasound (CUS) guided procedures stems from the displaced sense of hand-eye coordination that occurs when the operator looks away from the operating field to see the ultrasound display. The SF directly addresses many of these issues and therefore we believe that it is well suited for this application. We have already shown that novice US users learn vascular access procedures in training phantoms more quickly using the SF than CUS. We have also shown that IV team nurses already proficient in CUS guided PICC lines perform vascular access in training phantoms more quickly using the SF than CUS guidance. Finally, as mentioned earlier, we have shown that the SF can be used successfully to guide the placement of PICC lines. This study will test the hypothesis that the SF will successfully facilitate catheter placement in the subclavian, femoral, and internal jugular veins demonstrating equal vasculature visualization as conventional ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older
* The subjects will be patients already coming to interventional radiology services at University of Pittsburgh Medical Center (UPMC)-Presbyterian to have a CVA line placed.
* The racial, gender, and ethnic characteristics of the proposed subject population reflects the demographics of Pittsburgh and the surrounding area and/or the patient population of the University of Pittsburgh Medical Center.

Exclusion Criteria:

* Once 50 patients needing a particular insertion site have participated, no further recruiting will be done for patients needing the same insertion site.
* No exclusion criteria shall be based on race, ethnicity, gender, or HIV status.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Stetten, MD/PhD, Principal Investigator — University of Pittsburgh, Dept of Bioengineering
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States